CLINICAL TRIAL: NCT04649931
Title: Study to Evaluate Whether Differences in Exhaled Breath Can be Identified Using Ion Mobility Spectrometry (IMS) in Subjects Tested Positive for SARS-CoV-2 Infection and Subjects Tested Negative
Brief Title: Differences in Exhaled Breath by Using Ion Mobility Spectrometry (IMS) in Subjects Tested for SARS-CoV-2 Infection (COVID-19 Disease)
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Collaborators: CeGaT GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: HC-N-H-2006
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: SARS (Severe Acute Respiratory Syndrome); Covid19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — Ion Mobility Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ion Mobility Spectrometry (IMS) — Two breathing gas samples will be taken from each study participant using ion mobility spectrometry with an ultrasound-based spirometer. The total sampling time is 1 minute (at least 5-7 breath takes) following an analysis time of 5-12 minutes.

SUMMARY:
Breath gas analysis is the evaluation of exhaled breath. It aims to evaluate the volatile organic compounds (VOCs) in exhaled breath.

In this feasibility study it is intended to find specific peaks/pattern in exhaled breath indicating an infection with SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2).

ELIGIBILITY:
Inclusion Criteria:

* PCR (= Polymerase Chain Reaction) testing for SARS CoV-2 will be/has been performed in a timely manner of sampling exhaled breath or PCR test for SARS-CoV-2 was performed within 96 hours, but preferably within 48 hours before sampling exhaled breath and PCR test result is already available
* Subject must be able to comply with study-specific procedures, e.g.is able to comply with breathing commands

Exclusion Criteria:

* Previous (history) SARS-CoV-2 infection, independent of the current episode
* Participation in a therapeutic study prior to breath analysis which could influence the result of the breath analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected or diagnosed SARS-CoV-2 infection.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 related volatile organic compounds (VOC) | 1 hour after breath gas sampling

SECONDARY OUTCOMES:
To compare the SARS-CoV-2 specific VOC with the clinical symptoms of COVID-19 (Corona Virus Disease 2019) | within 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Schaefer, Prof. Dr., Principal Investigator — University Hospital Marburg, Zentrum für unerkannte und seltene Erkrankungen (ZusE)
Locations (1):
- University Hospital Gießen and Marburg (UKGM), site Marburg, Marburg, Germany